CLINICAL TRIAL: NCT01100034
Title: A LONG-TERM, PROSPECTIVE, OBSERVATIONAL COHORT STUDY OF THE SAFETY AND EFFECTIVENESS OF ETANERCEPT IN THE TREATMENT OF PAEDIATRIC PSORIASIS PATIENTS IN A NATURALISTIC SETTING: A POST-AUTHORISATION SAFETY STUDY (PASS)
Brief Title: Study Evaluating the Safety and Effectiveness of Etanercept for the Treatment of Pediatric Psoriasis
Acronym: PURPOSE
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881X1-4654; B1801035 (Other: Alias Study Number)
Record Dates: First submitted 2010-04-06; First posted 2010-04-08 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Psoriasis
Keywords: pediatric psoriasis; etanercept; PASS; safety; effectiveness
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: pediatric patients with plaque psoriasis on etanercept
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Expected duration of 24 weeks as one course
  Other Names: Enbrel

SUMMARY:
Psoriasis is a chronic, often severe, autoimmune condition that affects approximately 2% of the world's population. The epidemiology of pediatric psoriasis has not been well documented and no treatment guidelines exist for pediatric psoriasis.

Etanercept is a biologic drug and has been licensed for the treatment of chronic severe plaque psoriasis in children and adolescents (6-17 years of age) who are inadequately controlled by or are intolerant to, other systemic therapies or phototherapies. Although the long-term safety and efficacy of etanercept in children with juvenile idiopathic arthritis (JIA) has been studied and the short-term safety profile of etanercept in both JIA and pediatric psoriasis appears similar, there is limited data available about the long-term effects of etanercept in pediatric psoriasis, especially with respect to malignancy. The aim of this study is to assess the safety and effectiveness of etanercept for the treatment of pediatric psoriasis in Europe. Patients aged <=17 with plaque psoriasis diagnosed by a dermatologist will be invited to participate in the registry only after a clinical decision has been made to prescribe etanercept. The safety of the drug and how well the drug works will be evaluated during the follow-up period. The follow-up period will last 5 years and patients will be followed up every 3 months for the first 2 years and every 6 months for the next 3 years or until the end of study.

DETAILED DESCRIPTION:
Non-probability sample

ELIGIBILITY:
Inclusion Criteria:

* 17 years of age or younger
* Diagnosed with plaque psoriasis by a dermatologist.
* Prior to enrollment, there must be a clinical decision to initiate etanercept for the treatment of plaque psoriasis and etanercept must then be initiated.
* Actively being treated with etanercept, regardless of length of treatment prior to enrollment
* Willing to provide written informed consent

Exclusion Criteria:

* Prior therapy with any biologic agent other than etanercept
* History of malignancy

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: dermatology clinics
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2010-11-19 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- France (4):
  - Centre Hospitalier Victor Dupouy / Service de Dermatologie, Argenteuil
  - CHRU Tours Hopital Trousseau, Chambray-lès-Tours
  - CHU de Nantes - Hôtel Dieu, Nantes
  - CH Quimper Cornouaille, Quimper
- Germany (9):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Universitaetsklinik Koeln, Cologne
  - Universitaetsklinik Carl Gustav Carus, Dresden
  - Hautklinik Universitaetsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - J W Goethe Universitaet Frankfurt, Frankfurt am Main
  - Kath. Kinderkrankenhaus Wilhelmstift, Hamburg
  - Kinderklinik der Johannes-Gutenberg Universitat Mainz, Mainz
  - Asklepios Klinik Sankt Augustin GmbH, Sankt Augustin
- Greece (3):
  - Andreas Syngros Hospital, Athens
  - University of Athens, Andreas Syngros Hospital, Athens
  - Skin and Venereal Diseases' Hospital, Thessaloniki
- Heim Pal Children's Hospital, Budapest, Hungary
- Italy (6):
  - Universita degli Studi di Napoli Federico II, Napoli
  - Universita degli Studi di Napoli, Napoli
  - University of Padova, Padua
  - ARNAS Civico Di Gristina M Ascoli, Palermo
  - Università Cattolica del Sacro Cuore Policlinico A., Roma
  - Ospitale Alfredo Fiorini, Terracina
- Netherlands (2):
  - UMC St Radbound, Nijmegen
  - Erasmus MC, Rotterdam
- Hospital Santa Maria, Lisbon, Portugal
- Spain (3):
  - Hospital de la Santa Cruz y San Pablo, Barcelona
  - Hospital Parc Tauli, Barcelona
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881X1-4654&StudyName=Study%20Evaluating%20the%20Safety%20and%20Effectiveness%20of%20Etanercept%20for%20the%20Treatment%20of%20Pediatric%20Psoriasis

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Participants who were diagnosed with plaque psoriasis and on routine treatment of etanercept as per standard clinical practice were enrolled in this study and observed for approximately 5 years. Participants were observed for every 3 months during the first 2 years of the study and every 6 months thereafter for 3 years.
Period: Overall Study
Arm/Group | Etanercept
Started | 72
Completed | 29
Not Completed | 43
Not completed — Lost to Follow-up | 11
Not completed — Withdrawal of parent/guardian consent | 1
Not completed — Withdrawal by Subject | 4
Not completed — Sponsor decision | 21
Not completed — Participated in another clinical trial | 1
Not completed — Participants moved to another hospital | 4
Not completed — Site closed due to non-responsiveness | 1

BASELINE CHARACTERISTICS:
Population: Analysis population included all enrolled participants who were documented as having received at least 1 dose of etanercept.
Arm/Group | Etanercept
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.5 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — For Unknown: as per local regulations of France and Portugal, race/ethnicity should not be disclosed hence 11 participants from France and Portugal captured as Unknown.
  Participants
    White or Caucasian | 56
    Black | 1
    Other Asian | 2
    Other | 2
    Unknown | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Infections, Opportunistic Infections of Interest and Malignancies: Prospective Participants
Description: Serious infections were defined as any infections those were life-threatening or resulted in disability, infections requiring intravenous antibiotic treatment and hospitalisation. Opportunistic infections of interest included protocol-specified infections due to bacteria: Salmonella bacteremia, Campylobacteriosis, Shigellosis, Mycobacterium tuberculosis, Mycobacterium avium, Mycobacterium kansasii, Syphilis, Pseudomonas aeruginosa, Acinetobacter baumannii, Listeriosis, Nocardiosis, Legionellosis, Actinomycosis, Bartonellosis; Fungal: Aspergillosis, Invasive Candida albicans, Coccidioidomycosis, Cryptococcosis, Histoplasmosis, Blastomycosis, Paracoccidioidomycosis, Sporotrichosis, Penicilliosis, Zygomycosis and Pneumocystosis; Protozoans: Cryptosporidiosis, Isosporiasis, Microsporidiosis, Acanthamoebiasis, Toxoplasmosis, Trypanosomiasis and Leishmaniasis; Viral: Cytomegalovirus, John Cunningham Virus, Disseminated or central nervous system herpes zoster, Kaposi's sarcoma and BK virus.
Time Frame: Baseline up to 5 years
Population: Prospective Participants: participants who started etanercept within 30 days before the enrollment date or any time after enrollment date. This outcome measure was planned to be analyzed in prospective participants only.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 32
Participants
  Serious Infections | 0
  Opportunistic Infections of interest | 0
  Malignancies | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs): Prospective Participants
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline up to 28 days after last dose of study drug (up to 61 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 32
Participants
  Treatment emergent AEs | 26
  Treatment emergent SAEs | 3

3. Primary Outcome: Number of Participants Who Discontinued From Etanercept During Initial Treatment Period: Prospective Participants
Description: Initial treatment period is defined as the period during which participants received Etanercept treatment for a duration of at least 24 weeks.
Time Frame: Baseline up to 24 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 32
Participants | 3

4. Primary Outcome: Number of Participants Who Discontinued From Etanercept After Initial Treatment Period: Prospective Participants
Description: as for outcome 3
Time Frame: Week 24 up to Week 216
Population: Prospective Participants: participants who started etanercept within 30 days before the enrollment date or any time after enrollment date. This outcome measure was planned to be analyzed in prospective participants only. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 5
Participants | 4

5. Primary Outcome: Percentage of Participants Who Required Subsequent Treatment With Etanercept or Other Systemic Therapies After Completion of Initial Treatment Period: Prospective Participants
Description: Participants those who completed the initial treatment period of at least 24 weeks and entered the follow up period, and during the follow up period who required subsequent treatment with etanercept or other systemic therapies were reported.
Time Frame: Week 24 up to Week 216
Population: Prospective Participants: participants who started etanercept within 30 days before the enrollment date or any time after enrollment date. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies the participants evaluable at specific rows.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 28
percentage of participants
  Etanercept therapies | 17.9
  Other Systemic Therapies: number analyzed (Participants) | 15
  Other Systemic Therapies | 26.7

6. Secondary Outcome: Duration of Subsequent Etanercept Treatment After Completion of Initial Treatment Period
Time Frame: Week 24 up to Week 216
Population: Analysis population included all enrolled participants who were documented as having received at least 1 dose of etanercept. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Etanercept
Number analyzed (Participants) | 29
weeks | 146.3 (119.9)

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of study drug (up to 61 months)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both a serious and non-serious event during study.
Arm/Group | Etanercept
All-Cause Mortality (participants affected / at risk) | 0/72
Serious Adverse Events (participants affected / at risk) | 11/72
Other Adverse Events (participants affected / at risk) | 44/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=72)
Angina pectoris (Cardiac disorders) | 1
Drug ineffective (General disorders) | 2
Hepatic steatosis (Hepatobiliary disorders) | 1
Chronic tonsillitis (Infections and infestations) | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Paraesthesia (Nervous system disorders) | 1
Anorexia nervosa (Psychiatric disorders) | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=72)
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Conjunctivitis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Drug ineffective (General disorders) | 17
Injection site erythema (General disorders) | 1
Injection site pain (General disorders) | 1
Injection site reaction (General disorders) | 2
No adverse event (General disorders) | 1
Pyrexia (General disorders) | 1
Acute tonsillitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Ear infection (Infections and infestations) | 3
Eczema infected (Infections and infestations) | 1
Enterovirus infection (Infections and infestations) | 2
Gastroenteritis viral (Infections and infestations) | 2
Gastrointestinal infection (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 18
Otitis media (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 3
Rhinitis (Infections and infestations) | 1
Scarlet fever (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1
Sunburn (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Eosinophil count increased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Transient global amnesia (Nervous system disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2
Somatoform disorder neurologic (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 2
Vitiligo (Skin and subcutaneous tissue disorders) | 1
Venous thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/34/NCT01100034/SAP_000.pdf
  • Study Protocol (2014-07-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT01100034/Prot_001.pdf